CLINICAL TRIAL: NCT01975428
Title: Scripps Wired for Health Monitoring Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scripps Translational Science Institute (Other)
Collaborators: Scripps Health (Other)
Responsible Party: Principal Investigator, Eric Topol, MD, Director, Scripps Translational Science Institute, Scripps Translational Science Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Scripps WFH Study
Record Dates: First submitted 2012-10-17; First posted 2013-11-04 (Estimated); Results first posted 2021-07-07 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Diabetes; Hypertension; Cardiac Arrhythmia
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): All study participants, including participants randomized to the control arm, were enrolled in the HealthComp disease management program, which involved outreach by HealthComp nursing staff for purposes of relaying medical education and wellness information with regard to disease prevention and chronic disease management.
  Interventions: Behavioral: Control
- DM Pgm + device (Active Comparator): Disease management (DM) program plus a device corresponding to an individual's disease(s):
  iBGStar - iPhone enabled capillary blood glucose meter. Subjects test blood glucose up to 4 times per day, every day.
  Withings BP monitor - iPhone enabled home blood pressure monitor. Subjects test their blood pressure 2 times per day, up to 3 days per week.
  iPhone enabled Alive Cor ECG monitor. Participants take an ECG reading only when symptomatic.
  Interventions: Device: DM Pgm + device

INTERVENTIONS:
Device: DM Pgm + device — Disease management program plus a device corresponding to an individual's disease(s):
  iBGStar - iPhone enabled capillary blood glucose meter. Subjects test blood glucose up to 4 times per day, every day.
  Withings BP monitor - iPhone enabled home blood pressure monitor. Subjects test their blood pressure 2 times per day, up to 3 days per week.
  iPhone enabled Alive Cor ECG monitor. Participants take an ECG reading only when symptomatic.
  Arms: DM Pgm + device
Behavioral: Control — All study participants, including participants randomized to the control arm, were enrolled in the HealthComp disease management program, which involved outreach by HealthComp nursing staff for purposes of relaying medical education and wellness information with regard to disease prevention and chronic disease management.
  Arms: Control

SUMMARY:
People with chronic diseases such as diabetes, hypertension (high blood pressure) and cardiac (heart) arrhythmias tend to go to the doctor more often and have more tests done than those without those diseases. This can lead to increasing costs of healthcare and extra visits to doctors and healthcare facilities.

There are now medical devices that can be used at home to monitor blood sugar, blood pressure, heart rhythms as well as other measurements. There have been some studies which show that when people take their own health readings, they are better able to control their disease, stay healthier and go to the doctor less often. In order to participate in the study participants will have been diagnosed with 1 or more of the following: Diabetes, Hypertension, Cardiac Arrhythmias.

This study is designed to test those devices and see if they can help participants stay healthier through the recording and tracking of health measurements. Investigators will also be testing how easy it is to use these devices and whether or how easy it is to fit them in their daily schedule. Participants will be given an iPhone for use during the study and their recordings will be stored and displayed on the phone.

DETAILED DESCRIPTION:
The study will evaluate the impact of a "Wireless Monitoring" intervention for chronically ill individuals with diabetes, hypertension, and arrhythmias. This project utilizes the concept of 'hot-spotting' in that investigators will aim to target individuals with the highest health care needs, which investigators have defined to be patients with these diagnoses who showed the highest health care utilization rates over the previous 12-month period based on reimbursement data from a large health care third party administrator. Investigators aim to determine if wireless monitoring can reduce health care service utilization and thus health care costs for the small number of patients who spend the greatest number of health care dollars, thereby cutting the overall amount of health care spending dramatically.

Furthermore, investigators will be assessing whether or not access to health measurement data and the possibility of receiving feedback from a study staff member will increase the compliance of patients to their medication regimen, recommended diet and exercise. It is anticipated that armed with their own health data, these patients will be less likely to need acute care visits

Study participants will be employees of Scripps Health or dependents of employees covered with Scripps insurance, administered by third-party administrator, Health Comp. In addition, patients will be currently enrolled or willing to enroll in Health Comp's Disease Management program. Investigators predict that in addition to participation in the program, wireless monitoring will be associated with decreased inpatient health service utilization (hospital admissions, days of hospitalization) and decreased outpatient health service utilization (emergency department visits, need-based primary care clinic visits, and need-based specialty clinic visits). Investigators predict that these decreases will translate into significant reductions in health care costs for the treatment group relative to a control group and relative to pre-monitoring utilization rates.

ELIGIBILITY:
Inclusion Criteria:

1. Scripps Health insured employee or adult family member
2. Internet access and e-mail
3. Provide permission for study staff to access medical records
4. Participating in Health Comp Disease Management program or willingness to join
5. English speaking
6. Within the past 12 months, a history of billing insurance for diagnostic codes consistent with diabetes, hypertension, and/or cardiac arrhythmia
7. 18 years and older
8. Willingness to use wireless devices and study iPhone

Exclusion Criteria:

1. Employee of Scripps Clinic Medical Group
2. Related to or household sharing with another study participant (if there are two people or more in one household that are eligible, the member that has the highest utilization will be invited to join first)
3. Unwilling or unable to grant informed consent
4. Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2012-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric J Topol, MD, Principal Investigator — Scripps Translational Science Institute
Locations (1):
- Scripps Translational Science Institute, La Jolla, California, United States

REFERENCES:
- [Derived] Kim JY, Wineinger NE, Steinhubl SR. The Influence of Wireless Self-Monitoring Program on the Relationship Between Patient Activation and Health Behaviors, Medication Adherence, and Blood Pressure Levels in Hypertensive Patients: A Substudy of a Randomized Controlled Trial. J Med Internet Res. 2016 Jun 22;18(6):e116. doi: 10.2196/jmir.5429. PMID 27334418

RESULTS

PARTICIPANT FLOW:
Groups:
- Control: Disease Management Program
  This program involves periodic calls from a Health Comp staff member to see how a participant was feeling and if they were having any health problems.
- DM Pgm + Device: This program involves periodic calls from a Health Comp staff member to see how a participant was feeling and if they were having any health problems.
  iBGStar - iPhone enabled capillary blood glucose meter plus disease management program. Subjects test blood glucose up to 4 times per day, every day.
  iBG Star Blood Glucose Monitor: Participants will measure their blood glucose up to 4 times per day, every day.
  iphone enabled Alive Cor ECG monitor. Participants take an ECG reading only when symptomatic Alive Cor Portable ECG monitor: Portable electrocardiogram. Subjects will monitor their cardiac rhythms only when they have symptoms.
  Withings BP monitor - iPhone enabled home blood pressure monitor. Subjects test their blood pressure 2 times per day, up to 3 days per week.
  Withings Blood Pressure monitor: Home blood pressure monitor. Participants will measure their blood pressure 2 times per day up to 3 times per week.
Period: Overall Study
Arm/Group | Control | DM Pgm + Device
Started | 85 | 97
Completed | 65 | 83
Not Completed | 20 | 14
Not completed — Lost to Follow-up | 17 | 4
Not completed — Withdrawal by Subject | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- DM Pgm + Device: All study participants, including participants randomized to the control arm, were enrolled in the HealthComp disease management program, which involved outreach by HealthComp nursing staff for purposes of relaying medical education and wellness information with regard to disease prevention and chronic disease management.
  iBGStar - iPhone enabled capillary blood glucose meter plus disease management program. Subjects test blood glucose up to 4 times per day, every day.
  iBG Star Blood Glucose Monitor: Participants will measure their blood glucose up to 4 times per day, every day.
  iphone enabled Alive Cor ECG monitor. Participants take an ECG reading only when symptomatic Alive Cor Portable ECG monitor: Portable electrocardiogram. Subjects will monitor their cardiac rhythms only when they have symptoms.
  Withings BP monitor - iPhone enabled home blood pressure monitor. Subjects test their blood pressure 2 times per day, up to 3 days per week.
  Withings Blood Pressure monitor: Home blood pressure monitor. Participants will measure their blood pressure 2 times per day up to 3 times per week.
- Total: Total of all reporting groups
Arm/Group | Control | DM Pgm + Device | Total
Number analyzed (Participants) | 85 | 97 | 182
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 75 | 80 | 155
  >=65 years | 10 | 17 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.5 (9.8) | 56.0 (9.0) | 55.0 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 63 | 112
  Male | 36 | 34 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 10 | 14
  Not Hispanic or Latino | 76 | 86 | 162
  Unknown or Not Reported | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 9 | 6 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 6 | 10
  White | 62 | 73 | 135
  More than one race | 4 | 10 | 14
  Unknown or Not Reported | 5 | 1 | 6
Region of Enrollment [Number; unit: participants]
  United States | 85 | 97 | 182

OUTCOME MEASURES:

1. Primary Outcome: Participant Perceptions of Utility of Monitoring
Description: Multidimensional Health Locus of Control (Form C). Measure of the source of reinforcements for health-related behaviors: primarily internal, a matter of chance, or under the control of doctors, or other people. The scale includes 18 questions where responders indicate they strongly disagree(1), moderately disagree(2) slightly disagree(3) slightly agree(4) moderately agree(5) or strongly agree(6). Questions can be found here: https://nursing.vanderbilt.edu/projects/wallstonk/form_c.php. Subscale measures are summed over responses: questions 1, 6, 8, 12, 13, & 17 measure feeling of internal control (range 6-36); questions 2, 4, 9, 11, 15, 16 measure feeling of chance (range 6-36); questions 3, 5, 14 measure control of doctors (range 3-18); & questions 7, 10, & 18 measure control of others (range 3-18). Higher scores represent greater agreement with the questions that generally indicate greater feelings of more chance in one's health. Results presented using the 'Chance' subscale below.
Time Frame: Measure at Day 180.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Control | DM Pgm + Device
Number analyzed (Participants) | 65 | 65
Score on a scale | 13.4 (5.8) | 11.3 (5.3)

2. Secondary Outcome: Total Health Care Utilization and Costs.
Description: Total health care utilization and costs in USD.
Time Frame: Total billed over 180 days.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Control | DM Pgm + Device
Number analyzed (Participants) | 65 | 83
Units on a scale | 5596 (22187) | 6026 (21426)

ADVERSE EVENTS:
Groups:
- Control: This program involves periodic calls from a Health Comp staff member to see how a participant was feeling and if they were having any health problems.
Arm/Group | Control | DM Pgm + Device
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/97
Other Adverse Events (participants affected / at risk) | 0/85 | 0/97

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No